CLINICAL TRIAL: NCT06148220
Title: A Study of the Clinical Application of [18F]RCCB6 and [68Ga]Ga-NOTA-RCCB6 PET/CT Imaging in the Diagnosis of CD70-expressing Multiple Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-779
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Kidney Cancer; Lymphomas; Positron Emission Tomography
MeSH Terms: conditions — Kidney Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with renal cancer (Experimental): Intravenous injection of 3.7 MBq [0.1 mCi]/kg of [18F]RCCB6 or [68Ga]Ga-NOTA-RCCB6 in a single dose
  Interventions: Radiation: [18F]RCCB6 and [68Ga]Ga-NOTA-RCCB6 PET/CT imaging
- patients with lymphoma (Experimental): Intravenous injection of 3.7 MBq [0.1 mCi]/kg of [18F]RCCB6 or [68Ga]Ga-NOTA-RCCB6 in a single dose
  Interventions: Radiation: [18F]RCCB6 and [68Ga]Ga-NOTA-RCCB6 PET/CT imaging

INTERVENTIONS:
Radiation: [18F]RCCB6 and [68Ga]Ga-NOTA-RCCB6 PET/CT imaging — Intravenous injection of 3.7 MBq [0.1 mCi]/kg of [18F]RCCB6 or [68Ga]Ga-NOTA-RCCB6 in a single dose

SUMMARY:
The aim of this study was to establish and optimize the [18F]RCCB6 and [68Ga]Ga-NOTA-RCCB6 PET/CT imaging method, and its physiological and pathological distribution characteristics, on the basis of which the diagnostic efficacy of the above imaging agents in renal cancer (especially clear cell renal cell carcinoma) and lymphoma was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 65 years of age and of either sex.
2. Affected with renal cancer or lymphoma confirmed by puncture or surgical pathology.
3. Informed consent must be signed in writing by the subject or his/her legal guardian or caregiver.
4. Willingness and ability to cooperate with all programs of this study.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. Severe hepatic and renal insufficiency;
  2. Targeted therapy prior to radiotherapy or PET/CT scan. Renal function: serum creatinine less than or equal to the upper limit of the normal range;
  3. Liver function: bilirubin, AST(SGOT)/ALT(SGPT) less than or equal to the upper limit of the normal range.
  4. History of serious surgery in the last month.
  5. Those who have participated in other clinical trials during the same period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-13 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete PET imaging | 90mins from time of injection
  1. Establishment and optimization of imaging method for [18F]RCCB6 or [68Ga]Ga-NOTA-RCCB6 PET/CT imaging. 2. Evaluating the sensitivity and specificity of using [18F]RCCB6 or [68Ga]Ga-NOTA-RCCB6 PET/CT in diagnosing renal cell carcinoma (especially metastatic clear cell renal carcinoma) and lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China

REFERENCES:
- [Derived] Zhou X, Wu Q, Zhai W, Zhang Y, Wu Y, Cao M, Wang C, Guan Y, Liu J, Xie F, Wei W. CD70-Targeted Immuno-PET/CT Imaging of Clear Cell Renal Cell Carcinoma: A Translational Study. J Nucl Med. 2024 Dec 3;65(12):1891-1898. doi: 10.2967/jnumed.124.268509. PMID 39510586